CLINICAL TRIAL: NCT01956669
Title: A Phase II Study of Pazopanib GW786034, NSC# 737754 in Children, Adolescents and Young Adults With Refractory Solid Tumors
Brief Title: Pazopanib Paediatric Phase II Trial Children's Oncology Group (COG) in Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Children's Oncology Group (Network)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 116731; 2013-003595-12 (EudraCT Number); CPZP034X2203 (Other: Novartis)
Record Dates: First submitted 2013-08-01; First posted 2013-10-08 (Estimated); Results first posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-07

CONDITIONS: Solid Tumours
Keywords: VEGF; Pazopanib; Sarcoma; GW786034; Refractory Solid Tumors
MeSH Terms: conditions — Sarcoma | interventions — pazopanib

STUDY DESIGN:
Intervention Model Description: The study design included a hierarchical 2-stage tumor response assessment with each cohort independent from one other.
  * Cohort 1: rhabdomyosarcoma (RMS)
  * Cohort 2: non-rhabdomyosarcomatous soft tissue sarcoma (NRSTS)
  * Cohort 3: Ewing sarcoma/pPNET
  * Cohort 4: osteosarcoma
  * Cohort 5: measurable neuroblastoma (mNeuroblastoma)
  * Cohort 6: evaluable neuroblastoma (eNeuroblastma)
  * Cohort 7: hepatoblastoma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pazopanib (Experimental): All subjects were treated with pazopanib GW786034 tablets at a dose of 450 mg/m^2/dose or as a powder in suspension at a dose of 225 mg/m^2/dose. The maximum daily dose administered was to be 800 mg for the tablet and 400 mg for suspension. If 225 mg/m^2/dose was not tolerated (>=2 DLTs in 6 evaluable subjects), the dose for subjects who required suspension was reduced to 160 mg/m^2/dose. A cycle was defined as 28 days with no rest periods between cycles.
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — Pazopanib was supplied as a series of aqueous film-coated tablets containing 200 mg (oval-shaped, white, packaged in bottles containing 34 tablets each), and 400 mg (oval-shaped, white, packaged in bottles containing 68 tablets each). Pazopanib Powder for Oral Suspension was a white to slightly colour powder supplied to the clinical sites in amber glass (United State Pharmacopeia (USP) Type III) bottles with child-resistant closures. Each bottle contains 5 g of pazopanib.
  Other Names: GW786034

SUMMARY:
The study design was an open-label Phase II pediatric clinical study. The purpose of Study X2203 was to identify any efficacy signal in subjects with the disease subtypes under study, when treated with pazopanib monotherapy. Furthermore, it was to define the toxicities of pazopanib in children, as well as examine biological markers, e.g. cytokines and angiogenic factors, that could help further characterize any response of pazopanib in children. Pazopanib was administered as monotherapy in tablet and powder suspension formulations at daily doses of 450 mg/m2/dose or 225 mg/m2/dose, respectively. The first 6 enrolled subjects receiving oral suspension formulation were assessed for tolerability and extended PK sampling; and, only if pazopanib was tolerated, subsequent subjects were enrolled at the same starting dose with the suspension. Dose escalation was not permitted. For the tablet, a dosing nomogram was used based on the subject's BSA. Dose reduction was dependent upon the toxicity of pazopanib and disease status of the infants, toddlers, children, adolescents, and young adults. Subjects could be as young as 1 year-old infants to screen for enrollment. Subjects were assessed for initial response after 8 weeks of treatment prior to Cycle 3. A cycle was defined as 28 days of pazopanib treatment with no rest period between cycles. Treatment was administered continuously once daily. Treatment was to be discontinued if there was evidence of disease progression, unacceptable treatment-related toxicity, pregnancy. Histological classification was an important diagnostic inclusion in these subjects with a wide variety of refractory solid tumors, i.e. 7 different tumor types and each being a cohort.

DETAILED DESCRIPTION:
The study design included a hierarchical 2-stage tumor response assessment with each cohort independent from one other. First, an initial 10 subjects were enrolled into each cohort. In the event of ≥ 1 response in any of these initial subjects, an additional 10 subjects may be enrolled in that cohort to proceed. In the event of ≥ 3 responses, the agent was considered effective. However after end of-stage 1, study enrollment stopped due to insufficient antitumor activity. Subjects who discontinued study treatment were followed for survival status. The study was to continue accruing data and thus, remained open for approximately 1 year from Last Subject Last Visit (LSLV).

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects must be at least 1 and less than or equal to 18 years of age at the time of study entry.
* Patients must have had histologic verification of one of the malignancies listed below at original diagnosis or at relapse - a) Rhabdomyosarcoma, b) Non-rhabdomyosarcomatous Soft Tissue Sarcoma (including desmoplastic small round cell tumor), c) Ewing Sarcoma / Peripheral Primitive Neuroectodermal Tumor (PNET), d) Osteosarcoma, e) Neuroblastoma (Measurable), f) Neuroblastoma (Evaluable), g) Hepatoblastoma.
* Patient must have disease that has either relapsed or is refractory to prior therap
* Patients who will be receiving the tablet formulation must have a body surface area (BSA) >= 0.84 m^2 (square meter) at baseline.
* Patients must have radiographically measurable disease (with the exception of neuroblastoma), Measurable disease is defined as the presence of at least one lesion on magnetic resonance imaging (MRI) or computed tomography (CT) scan that can be accurately measured with the longest diameter a minimum of 10 mm in at least one dimension (CT scan slice thickness no greater than 5 mm).
* Patients with neuroblastoma who do not have measurable disease but have iodine-131 - meta-iodobenzylguanidine positive (MIBG+) evaluable disease are eligible.
* Patients must have a Lansky or Karnofsky performance status score of >= 50, corresponding to Eastern Cooperative Oncology Group (ECOG) categories 0, 1 or 2. Use Karnofsky for subjects >= 16 years of age and Lansky for subjects <= 16 years of age.
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.
* Patients must not have received myelosuppressive chemotherapy within 3 weeks of enrollment onto this study (6 weeks if prior nitrosourea).
* At least 7 days must have elapsed since the completion of therapy with a growth factor that supports platelet or white cell number or function. At least 14 days must have elapsed after receiving peg-filgrastim.
* At least 7 days must have elapsed since the completion of therapy with a biologic agent. For biologic agents that have known adverse events occurring beyond 7 days after administration, the period prior to enrollment must be extended beyond the time during which adverse events are known to occur.
* Subjects may have received bevacizumab, VEGF-Trap, or other VEGF blocking tyrosine kinase inhibitors, provided that they did not progress while receiving one of these agents. Subjects may not have previously received pazopanib.
* At least 21 days must have elapsed since the completion of the last dose of VEGF-Trap, and at least 7 days since a VEGF blocking tyrosine kinase inhibitor. Subjects must have recovered from any VEGF blocking drug-related toxicity (e.g., proteinuria).
* > = 21 days must have elapsed from infusion of last dose of antibody and toxicity related to prior antibody therapy must have recovered to Grade <= 1.
* Radiotherapy: >=2 weeks must have elapsed since local palliative radiotherapy (XRT) (small port); >=3 months must have elapsed if prior Traumatic Brain Injury (TBI), craniospinal XRT or if >=50% radiation of pelvis; >=6 weeks must have elapsed if other substantial bone marrow irradiation was given.
* No evidence of active graft versus host disease and >=2 months must have elapsed since transplant or rescue
* Adequate Bone Marrow Function defined as peripheral absolute neutrophil count (ANC) >=1000/ microlitre (µL), platelet count >= 75,000/µL (transfusion independent, defined as not receiving platelet transfusions within a 7 day period prior to enrollment); and hemoglobin >= 8.0 grams (g)/decilitre (dL), may receive red blood cell (RBC) transfusions. Subjects with bone marrow involvement will be eligible for study (provided they meet the criteria) but will not be evaluable for hematologic toxicity.
* Adequate Renal and Metabolic Function defined as creatinine clearance or radioisotope Glomerular filtration rate (GFR) >= 70 millilitre (mL)/ (min)/1.73 meter (m)^2 or A serum creatinine based on age/gender as follows, age 1 to < 2 years (male-0.6 milligrams (mg)/dL, female-0.6 mg/dL), age 2 to < 6 years (male-0.8 mg/dL, female-0.8 mg/dL), age 6 to < 10 years (male-1 mg/dL, female-1 mg/dL), age 10 to < 13 years (male-1.2 mg/dL, female-1.2 mg/dL), age 13 to < 16 years (male-1.5 mg/dL, female-1.4 mg/dL), age >= 16 years (male-1.7 mg/dL, female-1.4 mg/dL), urine creatinine ratio of <1 or a urinalysis that is negative for protein; or, 24-hour urine protein level < 1000 mg/dL, adequate thyroid function ,no more than Grade 1 abnormalities of potassium, calcium (confirmed by ionized calcium), magnesium and phosphorous.
* Adequate Liver Function defined as total bilirubin <=1.5 x upper limit of normal (ULN) for age, serum glutamic-pyruvic transaminase (SGPT) Alanine transaminase (ALT) <=2.5 x ULN (for the purpose of this study, the ULN for SGPT is 45 U/L), Serum albumin >=2 g/dL. Must not have active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones, liver metastases or otherwise stable chronic liver disease per investigator assessment). NOTE: Stable chronic liver disease should generally be defined by the absence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, oesophageal or gastric varices, persistent jaundice, or cirrhosis. No known positivity of hepatitis B surface antigen (HBsAg), or of positive hepatitis C antibody.
* Adequate Cardiac Function defined as shortening fraction of >=27% by echocardiogram (while not receiving medications for cardiac function), or ejection fraction of >= 50% by gated radionuclide study (while not receiving medications for cardiac function), the corrected QTc interval by Bazett's formula (QTcB) <450 milliseconds (msec), and must not have a history of myocardial infarction, severe or unstable angina, peripheral vascular disease or familial QTc prolongation.
* Adequate Blood Pressure Control defined as a blood pressure (BP) <= the 95th percentile for age, height, and gender measured, subjects on stable doses of no more than one anti-hypertensive medication, with a baseline BP <= 95th percentile for age, height and gender, will be eligible.
* Central Nervous System (CNS) Function defined as subjects with a known history of seizures must have well-controlled seizures and may not be receiving enzyme-inducing anti-convulsants, CNS toxicity <= Grade 2.
* Adequate Coagulation defined as prothrombin time (PT) and partial thromboplastin time (PTT) <= 1.2 x upper limit of normal and an international normalized ratio (INR) <= 1.2.

Key Exclusion Criteria:

* Pregnant or breast-feeding women are not eligible for this study due to risks of fetal and teratogenic adverse events as seen in animal/human studies. Negative pregnancy tests must be obtained in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method beginning at the signing of the informed consent until at least 2 weeks after the last dose of the study drug. The definition of adequate contraception will be based on the judgment of the principal investigator or a designated associate. Study drug may also potentially be secreted in milk and therefore breastfeeding women are excluded.

Males (including those who have had vasectomies) with partners who can become pregnant will need to use birth control while on this study, as will their partner. Men are advised to use condoms during sexual intercourse while on study drug and continue to use adequate contraception for at least 2 weeks after the last dose of protocol therapy.

* Patients requiring corticosteroids who have not been on a stable or decreasing dose of corticosteroid for the 7 days prior to enrollment are not eligible.
* Patients who are currently receiving another investigational drug are not eligible.
* Patients who are currently receiving other anti-cancer agents or radiation therapy are not eligible.
* Patients who are currently receiving more than one anti-hypertensive medication (Grade 3) or whose blood pressure is not well controlled are not eligible for study enrollment.
* Patients must not be on therapeutic anticoagulation (Warfarin [coumadin] and/or low molecular weight heparin are prohibited). Prophylactic anticoagulation (i.e. intraluminal heparin) of venous or arterial access devices is allowed.
* Patients receiving drugs with a known risk of torsades de pointes are not eligible.
* Patients who require thyroid replacement therapy are not eligible if they have not been receiving a stable replacement dose for at least 4 weeks prior to study enrollment.
* Patients who are unable to swallow tablets or liquid are not eligible.
* Patients who have an uncontrolled infection are not eligible.
* Patients will be excluded if any of the following are present, evidence of active bleeding, intratumoral hemorrhage, or bleeding diathesis; History (within 6 months prior to study enrollment) of arterial thromboembolic events, including transient ischemic attack (TIA) or cerebrovascular accident (CVA); history (within 6 months prior to study enrollment) of pulmonary embolism, deep venous thrombosis (DVT), or other venous thromboembolic event; history of clinically significant bleeding within 6 weeks prior to study enrollment.
* Patients with known involvement of the CNS by malignancy will be excluded.
* Patients who have had or are planning to have the following invasive procedures will be excluded- Major surgical procedure, laparoscopic procedure, open biopsy or significant traumatic injury within 28 days prior to Day 1 therapy (Subcutaneous port placement or central line placement is not considered major surgery but must be placed greater than 48 hours from planned Day 1 of therapy); Core biopsy within 7 days prior to Day 1 therapy; Fine needle aspirate or central line placement within 48 hours prior to Day 1therapy.
* Patients with serious or non-healing wound, ulcer, or bone fracture.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days of study enrollment.
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 57 (Actual)
Dates: Start 2014-10-08 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (31):
- United States (24):
  - Novartis Investigative Site, Long Beach, California
  - Novartis Investigative Site, Madera, California
  - Novartis Investigative Site, Orange, California
  - Novartis Investigative Site, Palo Alto, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Hartford, Connecticut
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, St. Petersburg, Florida
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Kansas City, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Hackensack, New Jersey
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Chapel Hill, North Carolina
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Fort Worth, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Norfolk, Virginia
  - Novartis Investigative Site, Seattle, Washington
- Canada (2):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Novartis Investigative Site, Prague, Czechia
- Novartis Investigative Site, Paris, France
- Novartis Investigative Site, Budapest, Hungary
- Novartis Investigative Site, Košice, Slovakia
- Novartis Investigative Site, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 30 centers in 7 countries: Canada (2), Czech Republic (1), France (1), Hungary (1), Slovakia (1), Spain (1) and USA (23).
Pre-assignment Details: 154 patients were planned to be enrolled in the study. A total of 57 patients were randomized and analyzed: cohort 1 (12), cohort 2 (11), cohort 3 (10), cohort 4 (10), cohort 5 (4), cohort 6 (4) and cohort 7 (6).
Groups:
- Cohort 1: Rhabdomyosarcoma (RMS); Cohort 2: Non-rhabdomyosarcomatous Soft Tissue Sarcoma (NRSTS); Cohort 3: Ewing Sarcoma/pPNET (Ewing); Cohort 4 (Osteosarcoma); Cohort 5: Measurable Neuroblastoma (mNeuroblastoma); Cohort 6: Evaluable Neuroblastoma (eNeuroblastma); Cohort 7 (Hepatoblastoma): Subjects were treated with pazopanib GW786034 tablets at a dose of 450 mg/m^2/dose or as a powder in suspension at a dose of 225 mg/m^2/dose. The maximum daily dose administered was to be 800 mg for the tablet and 400 mg for suspension. If 225 mg/m^2/dose was not tolerated (>=2 DLTs in 6 evaluable subjects), the dose for subjects who required suspension was reduced to 160 mg/m^2/dose. A cycle was defined as 28 days with no rest periods between cycles.
Period: Overall Study
Arm/Group | Cohort 1: Rhabdomyosarcoma (RMS) | Cohort 2: Non-rhabdomyosarcomatous Soft Tissue Sarcoma (NRSTS) | Cohort 3: Ewing Sarcoma/pPNET (Ewing) | Cohort 4 (Osteosarcoma) | Cohort 5: Measurable Neuroblastoma (mNeuroblastoma) | Cohort 6: Evaluable Neuroblastoma (eNeuroblastma) | Cohort 7 (Hepatoblastoma)
Started (All enrolled subjects who took 1 dose of medication included in mITT and Safety Sets) | 12 | 11 | 10 | 10 | 4 | 4 | 6
PK Set (All mITT subjects who had at least 1 PK sample analyzed) | 11 | 11 | 10 | 10 | 4 | 4 | 6
PKES Set (PK subset (received powder suspension and had at least 1 non-predose extended PK sampling)) | 4 | 0 | 3 | 0 | 1 | 1 | 5
Biomarker Set (All mITT subjects who had valid biomarker samples analyzed) | 12 | 11 | 9 | 9 | 3 | 4 | 3
Per Protocol Set (PP Set) | 9 | 10 | 6 | 9 | 4 | 4 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 12 | 11 | 10 | 10 | 4 | 4 | 6
Not completed — Disease Progression | 12 | 7 | 7 | 8 | 4 | 3 | 5
Not completed — Adverse Event | 0 | 2 | 2 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: modified Intent-to-treat (mITT) set comprised of all subjects who received at least one dose of protocol therapy
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Rhabdomyosarcoma (RMS) | Cohort 2: Non-rhabdomyosarcomatous Soft Tissue Sarcoma (NRSTS) | Cohort 3: Ewing Sarcoma/pPNET (Ewing) | Cohort 4 (Osteosarcoma) | Cohort 5: Measurable Neuroblastoma (mNeuroblastoma) | Cohort 6: Evaluable Neuroblastoma (eNeuroblastma) | Cohort 7 (Hepatoblastoma) | Total
Number analyzed (Participants) | 12 | 11 | 10 | 10 | 4 | 4 | 6 | 57
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.8 (3.82) | 15.7 (1.19) | 12.6 (4.67) | 14.1 (3.57) | 9.8 (5.91) | 13.0 (4.24) | 5.3 (4.80) | 11.9 (4.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 3 | 1 | 3 | 3 | 5 | 24
  Male | 7 | 7 | 7 | 9 | 1 | 1 | 1 | 33
Race/Ethnicity, Customized [Number; unit: Participants]
  White/Caucasian/European heritage | 9 | 7 | 6 | 7 | 3 | 3 | 1 | 36
  African American/African heritage | 1 | 2 | 3 | 2 | 0 | 1 | 1 | 10
  White Arabic/White North African heritage | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  American Indian/Alaskan native | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Central/South Asian heritage | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Japanese heritage | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Southeast Asian heritage | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian/other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Missing | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Objective Response Rate (ORR) in Subjects' With Tumors of Primary Interest (RMS, NRSTS or Ewing Sarcoma/pPNET)
Description: ORR was defined as the percentage of participants achieving either a Complete Response (CR) or partial Response (PR) based on the Investigator review. The responses were assessed by CT or MRI based on Response Evaluation Criteria In Solid Tumors Criteria (RECIST1.1). CR, disappearance of all target and non-target lesions; PR, at least a 30% decrease in the disease measurement, taking as reference the disease measurement done to confirm measurable disease at study enrollment, also no new lesion or progression of any non-target measurable lesion. Confirmation was based on the disease assessment at 1 cycle or at the next scheduled visit after the initial response. Only descriptive analysis performed.
Time Frame: From date of first dose of study treatment up to 55 months
Population: mITT Set
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1: Rhabdomyosarcoma (RMS) | Cohort 2: Non-rhabdomyosarcomatous Soft Tissue Sarcoma (NRSTS) | Cohort 3: Ewing Sarcoma/pPNET (Ewing)
Number analyzed (Participants) | 12 | 11 | 10
Percentage of Participants | 8.3 [0.4 to 33.9] | 0.0 [0.0 to 23.8] | 0.0 [0.0 to 25.9]

2. Secondary Outcome: Percentage of Participants Achieving Objective Response Rate (ORR) in Subjects' With Tumors of Secondary Interest (Osteosarcoma, mNeuroblastoma, eNeuroblastoma or Hepatoblastoma)
Description: ORR was defined as the percentage of participants achieving either a Complete Response (CR) or partial Response (PR) based on the Investigator review. For solid tumors with measurable diseases, such as osteosarcoma, the responses was based on RECIST1.1. CR, disappearance of all target and non target lesions; PR, at least a 30% decrease in the disease measurement, taking as reference the disease measurement done to confirm measurable disease at study enrollment, also no new lesion or progression of any non-target measurable lesion. For neuroblastoma with bone marrow response, morphology was determined by hematoxylin and eosin staining of the marrow and aspirates. For neuroblastoma MIBG+ only, the responses was assessed using Curie scale for lesion scoring; For hepatoblastoma, assessment may have included the serum AFP response, in addition to the RECIST1.1 methodology. Only descriptive analysis performed.
Time Frame: From date of first dose of study treatment up to 55 months
Population: mITT set
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 4 (Osteosarcoma) | Cohort 5: Measurable Neuroblastoma (mNeuroblastoma) | Cohort 6: Evaluable Neuroblastoma (eNeuroblastma) | Cohort 7 (Hepatoblastoma)
Number analyzed (Participants) | 10 | 4 | 4 | 6
Percentage of Participants | 0.0 [0.0 to 25.9] | 0.0 [0.0 to 52.7] | 0.0 [0.0 to 52.7] | 0.0 [0.0 to 39.3]

3. Secondary Outcome: Progression Free Survival (PFS) as Assessed by the Investigator by Cohort
Description: PFS was defined as the interval between the date of first dose of study medication and the earliest date of disease progression or death due to any cause. Disease progression was based on radiographic evidence, and assessments made by the investigator. According to RECIST1.1, disease progression was defined as at least a 20% increase in the sum of the disease measurements for measurable lesions, taking as reference the smallest disease measurement recorded since the start of treatment, or the appearance of one or more new lesions. For participants who did not progress or die, PFS was censored at the date of last adequate assessment or date of last adequate assessment prior to initiation of new anti-cancer therapy. Only descriptive analysis performed.
Time Frame: From date of first dose of study treatment up to 59 months
Population: mITT set
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Rhabdomyosarcoma (RMS) | Cohort 2: Non-rhabdomyosarcomatous Soft Tissue Sarcoma (NRSTS) | Cohort 3: Ewing Sarcoma/pPNET (Ewing) | Cohort 4 (Osteosarcoma) | Cohort 5: Measurable Neuroblastoma (mNeuroblastoma) | Cohort 6: Evaluable Neuroblastoma (eNeuroblastma) | Cohort 7 (Hepatoblastoma)
Number analyzed (Participants) | 12 | 11 | 10 | 10 | 4 | 4 | 6
Months | 1.8 [1.0 to 1.8] | 1.8 [0.3 to 13.8] | 2.3 [0.2 to 13.5] | 1.9 [0.5 to 5.3] | 4.9 [0.8 to 6.4] | 5.4 [3.6 to 24.4] | 1.8 [0.5 to 1.9]

4. Secondary Outcome: Time to Progression (TTP) by Cohort
Description: The TTP was defined as the interval between the date of first dose of protocol therapy and the earliest date of disease progression or death due to disease under study. Subjects were considered to have progressive disease if they had documented progression based on radiologic assessment as determined by investigator review. According to RECIST1.1, disease progression was defined as at least a 20% increase in the sum of the disease measurements for measurable lesions, taking as reference the smallest disease measurement recorded since the start of treatment, or the appearance of one or more new lesions. Only descriptive analysis performed.
Time Frame: From date of first dose of study treatment up to 59 months
Population: mITT set
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Rhabdomyosarcoma (RMS) | Cohort 2: Non-rhabdomyosarcomatous Soft Tissue Sarcoma (NRSTS) | Cohort 3: Ewing Sarcoma/pPNET (Ewing) | Cohort 4 (Osteosarcoma) | Cohort 5: Measurable Neuroblastoma (mNeuroblastoma) | Cohort 6: Evaluable Neuroblastoma (eNeuroblastma) | Cohort 7 (Hepatoblastoma)
Number analyzed (Participants) | 12 | 11 | 10 | 10 | 4 | 4 | 6
Months | 1.8 [1.0 to 1.8] | 1.8 [0.3 to 13.8] | 2.3 [0.2 to 13.5] | 1.9 [0.5 to 5.3] | 4.9 [0.8 to 6.4] | 14.9 [5.4 to 24.4] | 1.8 [0.5 to 1.9]

5. Secondary Outcome: Percentage of Participants Achieving Clinical Benefit Rate (CBR) by Cohort
Description: CBR was defined as the percentage of participants achieving either a confirmed complete response (CR) or confirmed partial response (PR) or Stable Disease (SD) for at least two protocol scheduled disease assessments based on RECIST1.1. CR, disappearance of all target and non-target lesions; PR, at least a 30% decrease in the disease measurement, taking as reference the disease measurement done to confirm measurable disease at study enrollment, also no new lesion or progression of any non-target measurable lesion; SD, neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease. Only descriptive analysis performed.
Time Frame: From date of first dose of study treatment up to 55 months
Population: mITT set
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1: Rhabdomyosarcoma (RMS) | Cohort 2: Non-rhabdomyosarcomatous Soft Tissue Sarcoma (NRSTS) | Cohort 3: Ewing Sarcoma/pPNET (Ewing) | Cohort 4 (Osteosarcoma) | Cohort 5: Measurable Neuroblastoma (mNeuroblastoma) | Cohort 6: Evaluable Neuroblastoma (eNeuroblastma) | Cohort 7 (Hepatoblastoma)
Number analyzed (Participants) | 12 | 11 | 10 | 10 | 4 | 4 | 6
Percentage of Participants | 8.3 [0.4 to 33.9] | 27.3 [7.9 to 56.4] | 20.0 [3.7 to 50.7] | 20.0 [3.7 to 50.7] | 50.0 [9.8 to 90.2] | 25.0 [1.3 to 75.1] | 0.0 [0.0 to 39.3]

6. Secondary Outcome: Duration of Response (DOR) by Cohort
Description: DoR was defined as the time from initial response to the first documented disease progression or death due to any cause, and was determined only for those participants from the mITT population with a confirmed response (CR or PR). Only descriptive analysis performed.
Time Frame: From date of first dose of study treatment up to 59 months
Population: mITT Set
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Rhabdomyosarcoma (RMS) | Cohort 2: Non-rhabdomyosarcomatous Soft Tissue Sarcoma (NRSTS) | Cohort 3: Ewing Sarcoma/pPNET (Ewing) | Cohort 4 (Osteosarcoma) | Cohort 5: Measurable Neuroblastoma (mNeuroblastoma) | Cohort 6: Evaluable Neuroblastoma (eNeuroblastma) | Cohort 7 (Hepatoblastoma)
Number analyzed (Participants) | 12 | 11 | 10 | 10 | 4 | 4 | 6
Months | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events

7. Secondary Outcome: Overall Survival (OS) by Cohort
Description: OS was defined as the time from the first dose of the study medication until death due to any cause. Only descriptive analysis performed.
Time Frame: From date of first dose of study treatment up to 61 months
Population: mITT Set
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Rhabdomyosarcoma (RMS) | Cohort 2: Non-rhabdomyosarcomatous Soft Tissue Sarcoma (NRSTS) | Cohort 3: Ewing Sarcoma/pPNET (Ewing) | Cohort 4 (Osteosarcoma) | Cohort 5: Measurable Neuroblastoma (mNeuroblastoma) | Cohort 6: Evaluable Neuroblastoma (eNeuroblastma) | Cohort 7 (Hepatoblastoma)
Number analyzed (Participants) | 12 | 11 | 10 | 10 | 4 | 4 | 6
Months | 5.6 [2.2 to 14.2] | 14.6 [1.5 to 20.1] | NA [4.3 to NA] — NA: Not estimable due to insufficient number of participants with events | 5.5 [1.5 to 7.0] | NA [2.6 to NA] — NA: Not estimable due to insufficient number of participants with events | 5.4 [3.6 to 24.4] | 5.7 [0.6 to NA] — NA: Not estimable due to insufficient number of participants with events

8. Secondary Outcome: Area Under the Plasma Concentration-time Curve Calculated From Time 0 to 8 h Postdose (AUC0-8h) and Calculated to the Last Quantifiable Concentration Point (AUClast) of Pazopanib by Cohort
Description: AUC0-8h and AUClast were calculated using a validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) and the LLOQ was 0.100 µg/mL. PK parameters were calculated from plasma concentration-time data using non-compartmental methods. Only descriptive analysis performed.
Time Frame: Day 1 of Cycle 1 (0, 0.5, 1, 2, 4, 6 and 8 hours post-dose); Cycle 1 Day 15 ± 1 day (0, 0.5, 1, 2, 4, 6 and 8 hours post-dose)
Population: PKES set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 1: Rhabdomyosarcoma (RMS) | Cohort 3: Ewing Sarcoma/pPNET (Ewing) | Cohort 5: Measurable Neuroblastoma (mNeuroblastoma) | Cohort 6: Evaluable Neuroblastoma (eNeuroblastma) | Cohort 7 (Hepatoblastoma)
Number analyzed (Participants) | 4 | 3 | 1 | 1 | 5
ng*hr/mL
  AUC0-8h (C1D1): number analyzed (Participants) | 2 | 2 | 0 | 0 | 3
  AUC0-8h (C1D1) | 195 (19.0) | 214 (93.2) |  |  | 135 (60.2)
  AUC0-8h (C1D15): number analyzed (Participants) | 4 | 2 | 1 | 1 | 5
  AUC0-8h (C1D15) | 388 (55.9) | 266 (36.1) | 475 (NA) — NA: Not estimable due to insufficient number of participants with events | 566 (NA) — NA: Not estimable due to insufficient number of participants with events | 229 (89.5)
  AUClast (C1D1): number analyzed (Participants) | 2 | 3 | 0 | 0 | 5
  AUClast (C1D1) | 194 (19.6) | 189 (65.8) |  |  | 135 (60.2)
  AUClast (C1D15): number analyzed (Participants) | 4 | 2 | 1 | 1 | 5
  AUClast (C1D15) | 966 (58.1) | 633 (35.4) | 1230 (NA) — NA: Not estimable due to insufficient number of participants with events | 1490 (NA) — NA: Not estimable due to insufficient number of participants with events | 607 (85.0)

9. Secondary Outcome: Observed Maximum Plasma Concentration (Cmax) of Pazopanib by Cohort
Description: Cmax was calculated using a validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) and the LLOQ was 0.100 µg/mL. PK parameters were calculated from plasma concentration-time data using non-compartmental methods. Only descriptive analysis performed.
Time Frame: as for outcome 8
Population: PKES set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1: Rhabdomyosarcoma (RMS) | Cohort 3: Ewing Sarcoma/pPNET (Ewing) | Cohort 5: Measurable Neuroblastoma (mNeuroblastoma) | Cohort 6: Evaluable Neuroblastoma (eNeuroblastma) | Cohort 7 (Hepatoblastoma)
Number analyzed (Participants) | 4 | 3 | 1 | 1 | 5
ng/mL
  Cmax (C1D1): number analyzed (Participants) | 4 | 3 | 1 | 0 | 5
  Cmax (C1D1) | 34.7 (14.7) | 35.6 (75.9) | 0.0 (NA) — NA: Not estimable due to insufficient number of participants with events |  | 22.4 (73.7)
  Cmax (C1D15): number analyzed (Participants) | 4 | 2 | 1 | 1 | 5
  Cmax (C1D15) | 56.7 (53.3) | 42.0 (42.3) | 69.6 (NA) — NA: Not estimable due to insufficient number of participants with events | 80.2 (NA) — NA: Not estimable due to insufficient number of participants with events | 33.4 (95.9)

10. Secondary Outcome: Time to Reach Peak or Maximum Concentration (Tmax) of Pazopanib by Cohort
Description: Tmax was calculated using a validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) and the LLOQ was 0.100 µg/mL. PK parameters were calculated from plasma concentration-time data using non-compartmental methods. Only descriptive analysis performed.
Time Frame: as for outcome 8
Population: PKES set
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1: Rhabdomyosarcoma (RMS) | Cohort 3: Ewing Sarcoma/pPNET (Ewing) | Cohort 5: Measurable Neuroblastoma (mNeuroblastoma) | Cohort 6: Evaluable Neuroblastoma (eNeuroblastma) | Cohort 7 (Hepatoblastoma)
Number analyzed (Participants) | 4 | 3 | 1 | 1 | 5
Hours
  Tmax (C1D1): number analyzed (Participants) | 4 | 3 | 1 | 0 | 5
  Tmax (C1D1) | 1 [0.00 to 2.00] | 2.02 [1.00 to 5.97] | 0.00 [0.00 to 0.00] |  | 2.00 [0.00 to 6.00]
  Tmax (C1D15): number analyzed (Participants) | 4 | 2 | 1 | 1 | 5
  Tmax (C1D15) | 2.50 [2.00 to 3.03] | 1.00 [1.00 to 1.00] | 3.47 [3.47 to 3.47] | 3.03 [3.03 to 3.03] | 3.00 [0.98 to 4.00]

11. Secondary Outcome: Pazopanib Steady-state Trough (Ctrough) Levels for Participants With Drug-related Grade 2 and Above Hypertension
Description: The relationship between toxicity (including hypertension) and pharmacokinetic parameters (pazopanib trough concentration) was analyzed. Only descriptive analysis performed.
Time Frame: From date of first dose of study treatment up to 61 months
Population: PK set. Only participants with a drug-related grade 2 and above hypertension event included in the analysis
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1: Rhabdomyosarcoma (RMS) | Cohort 2: Non-rhabdomyosarcomatous Soft Tissue Sarcoma (NRSTS) | Cohort 3: Ewing Sarcoma/pPNET (Ewing) | Cohort 4 (Osteosarcoma) | Cohort 5: Measurable Neuroblastoma (mNeuroblastoma) | Cohort 6: Evaluable Neuroblastoma (eNeuroblastma) | Cohort 7 (Hepatoblastoma)
Number analyzed (Participants) | 0 | 1 | 2 | 1 | 2 | 1 | 0
ng/mL |  | 97.1 (NA) — NA: Not estimable due to insufficient number of participants with events | 35.7 (22.6) | 35.7 (NA) — NA: Not estimable due to insufficient number of participants with events | 38.0 (20.8) | 63.7 (NA) — NA: Not estimable due to insufficient number of participants with events |

12. Secondary Outcome: Number of Participants With Genetic Alterations by Low and High Values of VEGFA and VEGFR1
Description: The frequency of genetic alterations observed in participants was presented by high and low baseline plasma levels for Vascular endothelial growth factor A (VEGF-A) and Vascular endothelial growth factor receptor 1 (VEGFR-1) biomarkers. The VEGFA and VEGFR1 levels above the median were classified as high and participants with median levels or below were classified as low. Only descriptive analysis performed for participants presenting with a genetic alteration.
Time Frame: predose Cycle 1 Day 1, Cycle 2 Day 1
Population: Biomarker set. Only participants with single nucleotide variant (SNV) were included in the analysis. The FLT1 gene was found to have a single SNV in one evaluable neuroblastoma participant.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Rhabdomyosarcoma (RMS) | Cohort 2: Non-rhabdomyosarcomatous Soft Tissue Sarcoma (NRSTS) | Cohort 3: Ewing Sarcoma/pPNET (Ewing) | Cohort 4 (Osteosarcoma) | Cohort 5: Measurable Neuroblastoma (mNeuroblastoma) | Cohort 6: Evaluable Neuroblastoma (eNeuroblastma) | Cohort 7 (Hepatoblastoma)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Participants
  VEGFA Low: VHL | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VEGFA Low: FLT1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  VEGFA Low: KDR | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VEGFA Low: HIF1A | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VEGFA Low: KRAS | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VEGFA Low: PIK3R1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VEGFA Low: MAPK1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VEGFA Low: PLCG1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VEGFA High: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VEGFA High: VHL | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VEGFA High: FLT1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VEGFA High: KDR | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VEGFA High: HIF1A | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VEGFA High: KRAS | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VEGFA High: PIK3R1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VEGFA High: MAPK1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VEGFA High: PLCG1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VEGFR1 Low: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VEGFR1 Low: VHL | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VEGFR1 Low: FLT1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VEGFR1 Low: KDR | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VEGFR1 Low: HIF1A | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VEGFR1 Low: KRAS | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VEGFR1 Low: PIK3R1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VEGFR1 Low: MAPK1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VEGFR1 Low: PLCG1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VEGFR1 High: VHL | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VEGFR1 High: FLT1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  VEGFR1 High: KDR | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VEGFR1 High: HIF1A | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VEGFR1 High: KRAS | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VEGFR1 High: PIK3R1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VEGFR1 High: MAPK1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VEGFR1 High: PLCG1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Summary for Plasma Biomarkers Levels on Cycle 1 Day 1 and Cycle 2 Day 1 by Cohort
Description: The following biomarker parameters were analyzed: proto-oncogene c-KIT (c-KIT), Fibroblast growth factor (FGF), Placental growth factor PGF), Angiopoietin-1 receptor (TIE2), Vascular endothelial growth factor A (VEGF-A), Vascular endothelial growth factor C (VEGF-C), Vascular endothelial growth factor D (VEGF-D), Vascular endothelial growth factor receptor 1 (VEGFR-1) and Vascular endothelial growth factor receptor 2 (VEGFR-2)). Only descriptive analysis performed.
Time Frame: predose Cycle 1 Day 1, Cycle 2 Day 1
Population: Biomarker set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram/milliliter (pg/mL)
Arm/Group | Cohort 1: Rhabdomyosarcoma (RMS) | Cohort 2: Non-rhabdomyosarcomatous Soft Tissue Sarcoma (NRSTS) | Cohort 3: Ewing Sarcoma/pPNET (Ewing) | Cohort 4 (Osteosarcoma) | Cohort 5: Measurable Neuroblastoma (mNeuroblastoma) | Cohort 6: Evaluable Neuroblastoma (eNeuroblastma) | Cohort 7 (Hepatoblastoma)
Number analyzed (Participants) | 12 | 11 | 9 | 9 | 3 | 4 | 3
picogram/milliliter (pg/mL)
  c-KIT (C1D1): number analyzed (Participants) | 12 | 10 | 9 | 8 | 2 | 3 | 3
  c-KIT (C1D1) | 139522.4 (29.4) | 142526.9 (24.3) | 135024.5 (25.9) | 137317.7 (23.9) | 142630.1 (18.0) | 113596.9 (26.6) | 119921.9 (30.6)
  c-KIT (C2D1): number analyzed (Participants) | 6 | 5 | 3 | 4 | 2 | 2 | 1
  c-KIT (C2D1) | 110154.0 (14.1) | 99962.7 (8.2) | 94307.1 (15.1) | 99989.6 (18.9) | 121497.7 (23.0) | 71216.5 (2.0) | 154558.2 (NA) — NA: Not estimable due to insufficient number of participants with events
  FGF (C1D1): number analyzed (Participants) | 3 | 3 | 2 | 2 | 0 | 1 | 0
  FGF (C1D1) | 7.8 (63.1) | 6.9 (71.1) | 8.3 (59.1) | 5.9 (6.0) |  | 13.5 (NA) — NA: Not estimable due to insufficient number of participants with events |
  FGF (C2D1): number analyzed (Participants) | 4 | 1 | 1 | 0 | 1 | 0 | 0
  FGF (C2D1) | 15.1 (68.9) | 6.2 (NA) — NA: Not estimable due to insufficient number of participants with events | 5.1 (NA) — NA: Not estimable due to insufficient number of participants with events |  | 6.6 (NA) — NA: Not estimable due to insufficient number of participants with events |  |
  PGF (C1D1): number analyzed (Participants) | 12 | 9 | 7 | 8 | 2 | 2 | 3
  PGF (C1D1) | 19.6 (245.7) | 8.9 (27.6) | 9.4 (36.9) | 10.5 (37.0) | 9.3 (6.2) | 13.7 (126.6) | 8.6 (29.7)
  PGF (C2D1): number analyzed (Participants) | 6 | 5 | 3 | 4 | 2 | 2 | 1
  PGF (C2D1) | 54.6 (259.4) | 27.8 (74.9) | 37.4 (82.9) | 63.2 (113.8) | 30.3 (300.5) | 225.2 (840.1) | 39.4 (NA) — NA: Not estimable due to insufficient number of participants with events
  TIE2 (C1D1): number analyzed (Participants) | 12 | 10 | 9 | 8 | 2 | 3 | 3
  TIE2 (C1D1) | 8086.8 (26.5) | 8180.0 (25.0) | 7280.6 (15.6) | 8574.9 (7.7) | 7439.8 (4.6) | 8179.2 (30.0) | 7842.2 (18.3)
  TIE2 (C2D1): number analyzed (Participants) | 6 | 5 | 3 | 4 | 2 | 2 | 1
  TIE2 (C2D1) | 8340.1 (11.5) | 7788.8 (11.5) | 7650.6 (22.7) | 7894.1 (17.4) | 8026.6 (28.2) | 6824.4 (32.0) | 8540.0 (NA) — NA: Not estimable due to insufficient number of participants with events
  VEGF-A (C1D1): number analyzed (Participants) | 12 | 10 | 9 | 8 | 2 | 3 | 3
  VEGF-A (C1D1) | 63.8 (133.8) | 46.1 (66.1) | 74.0 (98.0) | 82.9 (62.0) | 48.8 (39.0) | 62.2 (268.3) | 129.3 (46.6)
  VEGF-A (C2D1): number analyzed (Participants) | 6 | 5 | 3 | 4 | 2 | 2 | 1
  VEGF-A (C2D1) | 123.3 (140.6) | 77.2 (166.8) | 171.8 (126.0) | 179.4 (98.7) | 219.3 (40.4) | 1057.5 (750.0) | 208.9 (NA) — NA: Not estimable due to insufficient number of participants with events
  VEGF-C (C1D1): number analyzed (Participants) | 2 | 2 | 0 | 0 | 0 | 0 | 0
  VEGF-C (C1D1) | 121.4 (1.6) | 152.6 (84.7) |  |  |  |  |
  VEGF-C (C2D1): number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 0 | 0
  VEGF-C (C2D1) | 105.9 (NA) — NA: Not estimable due to insufficient number of participants with events | 339.9 (NA) — NA: Not estimable due to insufficient number of participants with events |  |  |  |  |
  VEGF-D (C1D1): number analyzed (Participants) | 12 | 10 | 9 | 8 | 2 | 3 | 3
  VEGF-D (C1D1) | 354.2 (54.6) | 372.3 (20.5) | 394.6 (21.6) | 375.4 (43.9) | 645.4 (108.7) | 351.7 (12.1) | 370.0 (75.9)
  VEGF-D (C2D1): number analyzed (Participants) | 6 | 5 | 3 | 4 | 2 | 2 | 1
  VEGF-D (C2D1) | 434.6 (77.4) | 501.8 (43.0) | 448.6 (16.9) | 551.7 (14.4) | 501.4 (50.1) | 791.4 (51.1) | 400.4 (NA) — NA: Not estimable due to insufficient number of participants with events
  VEGFR-1 (C1D1): number analyzed (Participants) | 12 | 10 | 9 | 8 | 2 | 3 | 3
  VEGFR-1 (C1D1) | 394.5 (292.3) | 175.7 (174.4) | 224.4 (121.7) | 134.6 (113.7) | 95.8 (42.9) | 367.5 (130.8) | 173.4 (109.6)
  VEGFR-1 (C2D1): number analyzed (Participants) | 6 | 5 | 3 | 4 | 2 | 2 | 1
  VEGFR-1 (C2D1) | 87.5 (98.5) | 534.3 (709.9) | 93.8 (121.1) | 140.0 (231.3) | 69.4 (4.9) | 76.4 (14.6) | 1811.6 (NA) — NA: Not estimable due to insufficient number of participants with events
  VEGFR-2 (C1D1): number analyzed (Participants) | 12 | 10 | 9 | 8 | 2 | 3 | 3
  VEGFR-2 (C1D1) | 31451.9 (22.6) | 31745.8 (20.6) | 33724.8 (15.8) | 34993.1 (17.6) | 31682.1 (12.1) | 39342.8 (14.7) | 30780.5 (6.0)
  VEGFR-2 (C2D1): number analyzed (Participants) | 6 | 5 | 3 | 4 | 2 | 2 | 1
  VEGFR-2 (C2D1) | 25099.6 (22.9) | 23059.9 (21.6) | 23502.8 (1.0) | 22154.3 (15.1) | 25385.9 (42.9) | 13621.6 (68.5) | 26266.9 (NA) — NA: Not estimable due to insufficient number of participants with events

14. Secondary Outcome: Summary for Change From Baseline Levels of Plasma Biomarkers by High and Low Pazopanib Steady State Trough Concentration and Cohort
Description: Participants with steady state trough concentration median levels for the following biomarker parameters (proto-oncogene c-KIT (c-KIT), Fibroblast growth factor (FGF), Placental growth factor PGF), Angiopoietin-1 receptor (TIE2), Vascular endothelial growth factor A (VEGF-A), Vascular endothelial growth factor C (VEGF-C), Vascular endothelial growth factor D (VEGF-D), Vascular endothelial growth factor receptor 1 (VEGFR-1) and Vascular endothelial growth factor receptor 2 (VEGFR-2)) above the median levels were classified as high or below median levels were classified as low. Only descriptive analysis performed.
Time Frame: predose Cycle 1 Day 1, Cycle 2 Day 1
Population: Biomarker set. Only patient with steady state trough plasma Pazopanib concentration included in the analysis.
Measure: Mean (Standard Deviation); unit: picogram/milliliter (pg/mL)
Arm/Group | Cohort 1: Rhabdomyosarcoma (RMS) | Cohort 2: Non-rhabdomyosarcomatous Soft Tissue Sarcoma (NRSTS) | Cohort 3: Ewing Sarcoma/pPNET (Ewing) | Cohort 4 (Osteosarcoma) | Cohort 5: Measurable Neuroblastoma (mNeuroblastoma) | Cohort 6: Evaluable Neuroblastoma (eNeuroblastma) | Cohort 7 (Hepatoblastoma)
Number analyzed (Participants) | 12 | 11 | 9 | 9 | 3 | 4 | 3
picogram/milliliter (pg/mL)
  c-KIT high trough concentration: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 1 | 0
  c-KIT high trough concentration |  |  | -76081.1 (NA) — NA: Not estimable due to insufficient number of participants with events | -40512.6 (NA) — NA: Not estimable due to insufficient number of participants with events |  | -51199.4 (NA) — NA: Not estimable due to insufficient number of participants with events |
  c-KIT low trough concentration: number analyzed (Participants) | 1 | 1 | 0 | 1 | 0 | 1 | 0
  c-KIT low trough concentration | -13480.5 (NA) — NA: Not estimable due to insufficient number of participants with events | -44973.7 (NA) — NA: Not estimable due to insufficient number of participants with events |  | -48764.1 (NA) — NA: Not estimable due to insufficient number of participants with events |  | -35678.6 (NA) — NA: Not estimable due to insufficient number of participants with events |
  FGF high trough concentration: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0
  FGF high trough concentration |  |  | -7.0 (NA) — NA: Not estimable due to insufficient number of participants with events |  |  |  |
  FGF low trough concentration: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PGF high trough concentration: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 1 | 0
  PGF high trough concentration |  |  | 78.3 (NA) — NA: Not estimable due to insufficient number of participants with events | 15.6 (NA) — NA: Not estimable due to insufficient number of participants with events |  | 45.4 (NA) — NA: Not estimable due to insufficient number of participants with events |
  PGF low trough concentration: number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 0 | 0
  PGF low trough concentration |  | 5.6 (NA) — NA: Not estimable due to insufficient number of participants with events |  | 28.3 (NA) — NA: Not estimable due to insufficient number of participants with events |  |  |
  TIE2 high trough concentration: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 1 | 0
  TIE2 high trough concentration |  |  | 2553.0 (NA) — NA: Not estimable due to insufficient number of participants with events | -509.4 (NA) — NA: Not estimable due to insufficient number of participants with events |  | -2708.2 (NA) — NA: Not estimable due to insufficient number of participants with events |
  TIE2 low trough concentration: number analyzed (Participants) | 1 | 1 | 0 | 1 | 0 | 1 | 0
  TIE2 low trough concentration | 1212.4 (NA) — NA: Not estimable due to insufficient number of participants with events | -1514.9 (NA) — NA: Not estimable due to insufficient number of participants with events |  | -918.4 (NA) — NA: Not estimable due to insufficient number of participants with events |  | -473.0 (NA) — NA: Not estimable due to insufficient number of participants with events |
  VEGF-A high trough concentration: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 1 | 0
  VEGF-A high trough concentration |  |  | 358.8 (NA) — NA: Not estimable due to insufficient number of participants with events | 34.3 (NA) — NA: Not estimable due to insufficient number of participants with events |  | -73.3 (NA) — NA: Not estimable due to insufficient number of participants with events |
  VEGF-A low trough concentration: number analyzed (Participants) | 1 | 1 | 0 | 1 | 0 | 1 | 0
  VEGF-A low trough concentration | 2436.6 (NA) — NA: Not estimable due to insufficient number of participants with events | 18.5 (NA) — NA: Not estimable due to insufficient number of participants with events |  | 52.3 (NA) — NA: Not estimable due to insufficient number of participants with events |  | 39.7 (NA) — NA: Not estimable due to insufficient number of participants with events |
  VEGF-C high trough concentration: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VEGF-C low trough concentration: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VEGF-D high trough concentration: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 1 | 0
  VEGF-D high trough concentration |  |  | 88.0 (NA) — NA: Not estimable due to insufficient number of participants with events | 139.7 (NA) — NA: Not estimable due to insufficient number of participants with events |  | 187.5 (NA) — NA: Not estimable due to insufficient number of participants with events |
  VEGF-D low trough concentration: number analyzed (Participants) | 1 | 1 | 0 | 1 | 0 | 1 | 0
  VEGF-D low trough concentration | 423.2 (NA) — NA: Not estimable due to insufficient number of participants with events | 44.1 (NA) — NA: Not estimable due to insufficient number of participants with events |  | 153.5 (NA) — NA: Not estimable due to insufficient number of participants with events |  | 90.8 (NA) — NA: Not estimable due to insufficient number of participants with events |
  VEGFR-1 high trough concentration: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 1 | 0
  VEGFR-1 high trough concentration |  |  | -217.5 (NA) — NA: Not estimable due to insufficient number of participants with events | 955.6 (NA) — NA: Not estimable due to insufficient number of participants with events |  | -49.7 (NA) — NA: Not estimable due to insufficient number of participants with events |
  VEGFR-1 low trough concentration: number analyzed (Participants) | 1 | 1 | 0 | 1 | 0 | 1 | 0
  VEGFR-1 low trough concentration | 484.1 (NA) — NA: Not estimable due to insufficient number of participants with events | -67.2 (NA) — NA: Not estimable due to insufficient number of participants with events |  | -7.7 (NA) — NA: Not estimable due to insufficient number of participants with events |  | -741.3 (NA) — NA: Not estimable due to insufficient number of participants with events |
  VEGFR-2 high trough concentration: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 1 | 0
  VEGFR-2 high trough concentration |  |  | -2620.0 (NA) — NA: Not estimable due to insufficient number of participants with events | -16136.9 (NA) — NA: Not estimable due to insufficient number of participants with events |  | -16838.7 (NA) — NA: Not estimable due to insufficient number of participants with events |
  VEGFR-2 low trough concentration: number analyzed (Participants) | 1 | 1 | 0 | 1 | 0 | 1 | 0
  VEGFR-2 low trough concentration | -12130.8 (NA) — NA: Not estimable due to insufficient number of participants with events | -7795.4 (NA) — NA: Not estimable due to insufficient number of participants with events |  | -8588.1 (NA) — NA: Not estimable due to insufficient number of participants with events |  | -10529.6 (NA) — NA: Not estimable due to insufficient number of participants with events |

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from first dose of study treatment plus 30 days post treatment, up to a maximum duration of 889 days.
Description: Any sign and symptom that occurs during the study treatment plus the 30 days post-treatment.
  Maximum exposure to study treatments = 889 days (cohort 1), 405 days (cohort 2), 404 days (cohort 3), 191 days (cohort 4), 196 days (cohort 5), 194 days (cohort 6) and 54 days (cohort 7).
Groups:
- Cohort 2: Nonrhabdomyosarcomatous Soft Tissue Sarcoma (NRSTS); Cohort 3: Ewing Sarcoma/pPNET (Ewing); Cohort 4 (Osteosarcoma); Cohort 5: Measurable Neuroblastoma (mNeuroblastoma); Cohort 6: Evaluable Neuroblastoma (eNeuroblastma); Cohort 7 (Hepatoblastoma); All Subjects: Subjects were treated with pazopanib GW786034 tablets at a dose of 450 mg/m^2/dose or as a powder in suspension at a dose of 225 mg/m^2/dose. The maximum daily dose administered was to be 800 mg for the tablet and 400 mg for suspension. If 225 mg/m^2/dose was not tolerated (>=2 DLTs in 6 evaluable subjects), the dose for subjects who required suspension was reduced to 160 mg/m^2/dose. A cycle was defined as 28 days with no rest periods between cycles.
Arm/Group | Cohort 1: Rhabdomyosarcoma (RMS) | Cohort 2: Nonrhabdomyosarcomatous Soft Tissue Sarcoma (NRSTS) | Cohort 3: Ewing Sarcoma/pPNET (Ewing) | Cohort 4 (Osteosarcoma) | Cohort 5: Measurable Neuroblastoma (mNeuroblastoma) | Cohort 6: Evaluable Neuroblastoma (eNeuroblastma) | Cohort 7 (Hepatoblastoma) | All Subjects
All-Cause Mortality (participants affected / at risk) | 3/12 | 0/11 | 1/10 | 3/10 | 0/4 | 1/4 | 1/6 | 9/57
Serious Adverse Events (participants affected / at risk) | 2/12 | 5/11 | 3/10 | 3/10 | 0/4 | 1/4 | 3/6 | 17/57
Other Adverse Events (participants affected / at risk) | 12/12 | 11/11 | 10/10 | 10/10 | 4/4 | 4/4 | 6/6 | 57/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Rhabdomyosarcoma (RMS) (N=12) | Cohort 2: Nonrhabdomyosarcomatous Soft Tissue Sarcoma (NRSTS) (N=11) | Cohort 3: Ewing Sarcoma/pPNET (Ewing) (N=10) | Cohort 4 (Osteosarcoma) (N=10) | Cohort 5: Measurable Neuroblastoma (mNeuroblastoma) (N=4) | Cohort 6: Evaluable Neuroblastoma (eNeuroblastma) (N=4) | Cohort 7 (Hepatoblastoma) (N=6) | All Subjects (N=57)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Wound infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Intracranial pressure increased (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Rhabdomyosarcoma (RMS) (N=12) | Cohort 2: Nonrhabdomyosarcomatous Soft Tissue Sarcoma (NRSTS) (N=11) | Cohort 3: Ewing Sarcoma/pPNET (Ewing) (N=10) | Cohort 4 (Osteosarcoma) (N=10) | Cohort 5: Measurable Neuroblastoma (mNeuroblastoma) (N=4) | Cohort 6: Evaluable Neuroblastoma (eNeuroblastma) (N=4) | Cohort 7 (Hepatoblastoma) (N=6) | All Subjects (N=57)
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 0 | 3 | 2 | 1 | 2 | 12
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 2 | 0 | 1 | 0 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 3
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deafness bilateral (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypothyroidism (Endocrine disorders) | 2 | 2 | 3 | 2 | 0 | 2 | 0 | 11
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Erythema of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Eye pain (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Eyelash discolouration (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Vision blurred (Eye disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 4
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 4 | 1 | 4 | 2 | 1 | 2 | 19
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 8
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 4 | 2 | 2 | 2 | 1 | 17
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 1 | 5 | 3 | 2 | 2 | 3 | 20
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 8 | 0 | 2 | 3 | 2 | 1 | 4 | 20
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Fatigue (General disorders) | 4 | 3 | 4 | 2 | 0 | 2 | 2 | 17
Feeling jittery (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Influenza like illness (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Nodule (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 3
Oedema peripheral (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Pain (General disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 4
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 5 | 1 | 2 | 3 | 1 | 0 | 4 | 16
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Otitis media acute (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 4
Urinary tract infection (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 4
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 5
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Tongue injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Alanine aminotransferase increased (Investigations) | 3 | 0 | 3 | 4 | 0 | 1 | 3 | 14
Amylase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 3
Aspartate aminotransferase increased (Investigations) | 4 | 0 | 3 | 3 | 1 | 1 | 4 | 16
Blood alkaline phosphatase (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 4
Blood creatinine increased (Investigations) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 3
Blood thyroid stimulating hormone increased (Investigations) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 3
Blood urea increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Carbon dioxide decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac murmur (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Creatinine urine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 3
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 4
Haemoglobin increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 3
Lymphocyte count decreased (Investigations) | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 5
Lymphocyte count increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Monocyte count increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 2 | 1 | 2 | 1 | 0 | 2 | 10
Platelet count decreased (Investigations) | 4 | 1 | 2 | 5 | 1 | 1 | 2 | 16
Protein total increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Red blood cell count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urine analysis abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Vanillyl mandelic acid urine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 1 | 2 | 1 | 0 | 1 | 2 | 7
White blood cell count decreased (Investigations) | 3 | 0 | 0 | 5 | 2 | 0 | 3 | 13
Decreased appetite (Metabolism and nutrition disorders) | 4 | 4 | 4 | 4 | 1 | 2 | 3 | 22
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 2 | 0 | 0 | 2 | 7
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 2 | 0 | 1 | 0 | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 4
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 5 | 2 | 2 | 0 | 1 | 16
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 4
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2 | 4 | 1 | 1 | 1 | 14
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 3 | 0 | 1 | 0 | 6
Dysgeusia (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 3
Headache (Nervous system disorders) | 2 | 3 | 2 | 2 | 1 | 0 | 1 | 11
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 3
Depression (Psychiatric disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 3
Insomnia (Psychiatric disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 3
Intentional self-injury (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Bladder pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Haematuria (Renal and urinary disorders) | 2 | 1 | 1 | 1 | 1 | 1 | 0 | 7
Haemoglobinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 4 | 1 | 2 | 3 | 1 | 1 | 1 | 13
Amenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Genital pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 3 | 3 | 0 | 1 | 1 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 2 | 1 | 1 | 0 | 7
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2 | 2 | 0 | 1 | 0 | 8
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 5
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hair colour changes (Skin and subcutaneous tissue disorders) | 1 | 2 | 3 | 2 | 1 | 3 | 1 | 13
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Macule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 3
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Skin depigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 3
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 2 | 2 | 4 | 1 | 1 | 2 | 13
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-05-23): https://cdn.clinicaltrials.gov/large-docs/69/NCT01956669/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-24): https://cdn.clinicaltrials.gov/large-docs/69/NCT01956669/SAP_001.pdf